CLINICAL TRIAL: NCT04201769
Title: A Standard Regimen of Dexamethasone in Comparison to Two Dex-sparing Regimens in Addition to NEPA in Preventing CINV in naïve NSCLC Patients to be Treated With Cisplatin Based Chemotherapy: a Three-arm, Open-label, Randomized Study
Brief Title: Dexamethasone-sparing Approach Including NEPA Against Emesis Caused by Cisplatin
Acronym: LUNG-NEPA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LUNG-NEPA
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: nausea; vomiting; lung cancer; DEX-Sparing
MeSH Terms: conditions — Vomiting; Nausea; Lung Neoplasms | interventions — netupitant, palosentron drug combination; netupitant; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase III, multicenter, randomized, open-label, parallel-group, active-comparator, three-arm, non-inferiority study
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): Oral Netupitant/Palonosetron (NEPA) and intravenous Dexamethasone (DEX) on Day 1 of chemotherapy.
  No further anti-emetic prophylaxis on days 2 thorough 4.
  Interventions: Drug: Netupitant/Palonosetron; Drug: Dexamethasone
- Arm B (Experimental): Oral Netupitant/Palonosetron (NEPA) and intravenous Dexamethasone (DEX) on Day 1 of chemotherapy.
  Oral dexamethasone 4 mg once per day in the morning of days 2 and 3.
  Interventions: Drug: Netupitant/Palonosetron; Drug: Dexamethasone
- Arm C (Active Comparator): Oral Netupitant/Palonosetron (NEPA) and intravenous Dexamethasone (DEX) on Day 1 of chemotherapy.
  Oral dexamethasone 4 mg twice per day on days 2 thorough 4.
  Interventions: Drug: Netupitant/Palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Netupitant/Palonosetron — NEPA is adiministered 60 minutes before chemotherapy, on day 1
  Other Names: Netupitant/Palonosetron 300-0.5 milligrams Oral Capsule [AKYNZEO]
Drug: Dexamethasone — Intravenous dexamethasone 12 mg is administered 30 minutes before chemotherapy initiation, on day 1.
  The administration of DEX in the subsequent days (2-4) depends on the randomly assignement to treatment arm

SUMMARY:
This study evaluates the possibility to reduce the total dose of dexamethasone, when administered with NEPA, to prevent chemotherapy-induced nausea and vomiting (CINV) in Non-Small Cell Lung Cancer (NSCLC) patients receiving a cisplatin-based chemotherapy

DETAILED DESCRIPTION:
On day 1 (day of chemotherapy), all eligible patients will receive oral NEPA (300 mg netupitant/0.5 mg palonosetron), 60 minutes before chemotherapy, and intravenous dexamethasone 12 mg, 30 minutes before chemotherapy initiation.

For the prevention of delayed CINV, patients will be assigned randomly to one of the following treatment arms:

* Test arm A: no further anti-emetic prophylaxis on days 2 thorough 4;
* Test arm B: oral dexamethasone 4 mg once per day in the morning of days 2 and 3;
* Reference arm C: oral dexamethasone 4 mg twice per day on days 2 thorough 4.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* Histologically or cytologically confirmed diagnosis of NSCLC
* Patients naїve to cisplatin-containing chemotherapy as well as any prior chemotherapy containing either highly or moderately emetogenic agents given for NSCLC or other malignancy.
* Patients scheduled to receive their first cycle of cisplatin-based chemotherapy at a dose ≥70 mg/m2 either alone or in combination with other agents of low or minimal potential of emetogenicity (i.e., pemetrexed, gemcitabine±bevacizumab, vinorelbine) as neo-adjuvant, adjuvant or palliative therapy. Patients with progressive disease on therapy with an EGFR-TKI (Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitors) and scheduled to receive cisplatin-based chemotherapy will be eligible for the study.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-1.
* Body Mass Index ≥18.5.
* Written informed consent before study entry.
* If women of childbearing potential age: effective contraceptive measures must be used during all the planned course of chemotherapy and up to 30 days after last NEPA administration.
* Normal hepatic function (≤2 times the upper limit of normal for liver transaminases) and renal function (creatinine ≤ 1.5 times the upper limit of normal).
* Ability and willingness of the patient to complete the diary and study questionnaires.

Exclusion Criteria:

* Symptomatic brain metastases.
* Patients scheduled to receive radiation therapy to the abdomen or pelvis within 1 week before day 1 or between day 1 and 5 following the first cycle of chemotherapy.
* Patients scheduled to receive concurrent chemo/radiotherapy for NSCLC.
* Treatment with investigational medications within 30 days before the study medication.
* Myocardial infarction within the last 6 months.
* Documented or known hypersensitivity to 5HT3RA (5-Hydroxytryptamine Receptor 3 Antagonists) or NK-1RA (Neurokinin-1 Receptor Antagonist) and excipients (see section 6.1 of Akynzeo SPC).
* Uncontrolled diabetes mellitus or active infection.
* Nausea and vomiting in the 24 hours before study treatment.
* Chronic use of systemic corticosteroids (except for topical and inhaled corticosteroids) or any other agent with anti-emetic potential. Patients receiving dexamethasone on the day before chemotherapy for prevention of the pemetrexed-induced skin rash will be eligible for the study.
* Patient's inability to take oral medication.
* Gastrointestinal obstruction or active peptic ulcer.
* Pregnancy or breast feeding.
* Prior malignancies at other sites except surgically treated non-melanoma skin cancer, superficial cervical cancer, or other cancer from which the patient had been disease-free for at least 5 years (see also inclusion criteria if prior chemotherapy treatment).
* Psychiatric or CNS (Central Nervous System) disorders interfering with ability to comply with study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | During the overall phase (day 1 thorough 5) of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  The proportion of patients achieving a complete response, defined as no emetic episode and no use of rescue medication, during the overall study period (day 1 thorough 5) of the first cycle of chemotherapy.

SECONDARY OUTCOMES:
CR (acute and delayed). | During the acute (within 24 hours post-chemotherapy) and delayed (days 2 thorough 5) phases of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  No emetic episode and no use of rescue medication, during the acute and delayed phases
Complete control | During the acute (within 24 hours post-chemotherapy), delayed (days 2 thorough 5) and overall (days 1 thorough 5) phases of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  No emetic episode, no rescue medication, and no more than mild nausea. Severity of nausea will be self-reported by the patient using a verbal scale (none, mild, moderate, and severe).
Proportion of patients with no emetic episode | During the acute (within 24 hours post-chemotherapy), delayed (days 2 thorough 5) and overall (days 1 thorough 5) phases of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  No emetic episode
Proportion of patients with no nausea | During the acute (within 24 hours post-chemotherapy), delayed (days 2 thorough 5) and overall (days 1 thorough 5) phases of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  No nausea. Severity of nausea will be self-reported by the patient using a verbal scale (none, mild, moderate, and severe).
Impact of nausea and vomiting on patient's quality of life | On day 6 of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  Impact of nausea and vomiting on patient's quality of life as recorded by the Italian version of the FLIE (Functional Living Index-Emesis) questionnaire, according to subjective assessment by each patient on day 6.
  The questionnaire consists of 18 questions: the first set of 9 questions refers to nausea and the second set of 9 questions refers to vomiting.
  Each question uses a visual analogue scale. Scale ranges are 1-7 (in some questions 1 indicates no effect on patient's quality of life, in other questions 1 indicates a great deal of an effect on patient's quality of life).
Patient global satisfaction with anti-emetic therapy, | On day 6 of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  Patient global satisfaction with antiemetic therapy, as measured by a Visual Analogue Scale (VAS) on day 6. Scale ranges are 0-10 (0 represents maximum dissatisfaction, 10 represents maximum satisfaction)
Safety profile | During all the safety study period (up to three weeks after the start of cisplatin-based chemotherapy)
  Safety profile according to NCI-CTCAE version 5.0
Cross-sectional baseline evaluation of weight loss (WL) | During the Screening phase (up to 7 days before the first cycle of chemotherapy administration - each cycle is 7 or 21 days)
  Weight loss will be assessed through the BMI (Body Mass Index) adjusted weight loss grading system (WLGS).
  WL as classified according to WLGS, a grading system using the combination of %WL and BMI categories. The analysis will be laid out in a 5x5 matrix representing five different %WL categories within each of the five different BMI categories (25 possible combinations of WL and BMI).
  Percentage of WL will be defined as follows: [(current weight in Kg - previous weight in Kg)/previous weight in Kg] x 100. Previous patient weight (i.e., the usual weight) within the last 6 months (or "usual weight") will be also collected at baseline. BMI will be calculated as current weight/square of the body height (Kg/m2);
Nutritional intake | During the Screening phase (up to 7 days before the first cycle of chemotherapy administration - each cycle is 7 or 21 days)
  Nutritional intake will be assessed with an ad hoc question adapted from the Patient Generated-Subjective Global Assessment (PG-SGA) questionnaire.
Cancer-related symptom self-assessment | On day 1 of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  Cancer-related symptom self-assessment, as recorded by the Italian version of the ESAS (Edmonton Symptom Assessment Scale) questionnaire, according to subjective assessment by each patient on day 1 (before cisplatin-based chemotherapy initiation), will be performed.
  The ESAS is a validated symptom inventory tool assessing the current intensity of 10 common symptoms in cancer patients, each with an 11-point numerical rating scale from 0 (no symptom) to 10 (worst intensity).
Cancer-related symptom self-assessment association with WLGS and nutritional intake | On day 1 of the first cycle of cisplatin-based chemotherapy (each cycle is 7 or 21 days)
  The association between Cancer-related symptom self-assessment and WLGS and nutritional intake will be examined using linear regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Bria, MD, Study Chair — Fondazione Policlinico Universitario "A. Gemelli" IRCCS, UCSC - Rome (Italy); Luigi Celio, MD, Study Director — Fondazione IRCCS "Istituto Nazionale Tumori" - Milan (Italy)
Locations (26):
- Italy (26):
  - ASST Bergamo Ovest - Ospedale di Teviglio, Treviglio, BG
  - Azienda ULSS 1 Dolomiti - Ospedale Santa Maria del Prato, Feltre, BL
  - ASST Ovest Milanese - Ospedale di Legnano, Legnano, MI
  - AOU San Luigi Gonzaga, Orbassano, TO
  - A.O.U. Consorziale Policlinico di Bari, Bari
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Cosenza, Cosenza
  - ASST Lecco - P.O. "A. Manzoni", Lecco
  - A.O.U. Policlinico di Modena, Modena
  - Ospedale San Gerardo - ASST Monza, Monza
  - A.O.R.N. dei Colli - Ospedale Monaldi, Napoli
  - Casa di Cura di Alta Specialità Dip. Oncologico di III livello "La Maddalena", Palermo
  - Ospedale S. Maria della Misericordia, Perugia
  - Ospedale di Piacenza, Piacenza
  - IRCCS Arcispedale S. Maria Nuova, Reggio Emilia
  - A.O. San Camillo Forlanini, Roma
  - A.O. San Giovanni - Addolorata, Roma
  - Fondazione Policlinico "A. Gemelli" - Università Cattolica Sacro Cuore, Roma
  - Istituto Nazionale Tumori "Regina Elena", Roma
  - Policlinico Tor Vergata, Roma
  - Ospedale Civile SS. Annunziata, Sassari
  - Ospedale Umberto I - RAO SR, Syracuse
  - P.O. "San Giuseppe Moscati", Taranto
  - Azienda ULSS 2 Marca Trevigiana - Ospedale di Treviso, Treviso
  - A.O.U.I. Verona - Policlinico "G.B. Rossi", Verona

REFERENCES:
- [Derived] Celio L, Aapro M. Characteristics of nausea and its impact on health-related quality of life in cisplatin-treated patients receiving dexamethasone-sparing prophylaxis: an analysis of the LUNG-NEPA study. Support Care Cancer. 2024 Mar 4;32(3):204. doi: 10.1007/s00520-024-08406-5. PMID 38433125
- [Derived] Celio L, Bartsch R, Aapro M. Dexamethasone-sparing regimens with NEPA (netupitant/palonosetron) for the prevention of chemotherapy-induced nausea and vomiting in older patients (>65 years) fit for cisplatin: A sub-analysis from a phase 3 study. J Geriatr Oncol. 2023 Jul;14(6):101537. doi: 10.1016/j.jgo.2023.101537. Epub 2023 Jun 7. PMID 37290207
- [Derived] Celio L, Cortinovis D, Cogoni AA, Cavanna L, Martelli O, Carnio S, Collova E, Bertolini F, Petrelli F, Cassano A, Chiari R, Zanelli F, Pisconti S, Vittimberga I, Letizia A, Misino A, Gernone A, Bonizzoni E, Pilotto S, De Placido S, Bria E. Exploratory analysis of the effect of a dexamethasone-sparing regimen for prophylaxis of cisplatin-induced emesis on food intake (LUNG-NEPA study). Sci Rep. 2023 Jan 23;13(1):1257. doi: 10.1038/s41598-023-28464-9. PMID 36690734
- [Derived] Celio L, Cortinovis D, Cogoni AA, Cavanna L, Martelli O, Carnio S, Collova E, Bertolini F, Petrelli F, Cassano A, Chiari R, Zanelli F, Pisconti S, Vittimberga I, Letizia A, Misino A, Gernone A, Bonizzoni E, Pilotto S, De Placido S, Bria E. Evaluating the impact of chemotherapy-induced nausea and vomiting on daily functioning in patients receiving dexamethasone-sparing antiemetic regimens with NEPA (netupitant/palonosetron) in the cisplatin setting: results from a randomized phase 3 study. BMC Cancer. 2022 Aug 24;22(1):915. doi: 10.1186/s12885-022-10018-3. PMID 35999527